CLINICAL TRIAL: NCT05109910
Title: Prospective Randomized Controlled Trial To Evaluate The Prognostic Role of Lymph Node Dissection In Men With Prostate Cancer Treated With Radical Prostatectomy
Brief Title: The Prognostic Role of Lymph Node Dissection In Men With Prostate Cancer Treated With Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20PRD
Record Dates: First submitted 2021-08-26; First posted 2021-11-05 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Lymph node dissection; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical prostatectomy with an extended pelvic lymph node dissection (Active Comparator): According to the standard of care, patients in this arm will receive a radical prostatectomy with a standard bilateral ePLND. This includes the removal of lymph nodes within the obturator fossa and bilateral to the external iliac artery, internal iliac artery and common iliac artery up to the ureteral-vessel crossing.
  Interventions: Procedure: Pelvic lymph node dissection
- Radical prostatectomy without an extended pelvic lymph node dissection (No Intervention): Patients in this arm will undergo a radical prostatectomy without a bilateral extended pelvic lymph node dissection. In case of intraoperatively found suspicious lymph nodes, a lymphadenectomy is performed. According to the intention to treat principle, patients with intraoperatively removed lymph nodes remain included in the study.

INTERVENTIONS:
Procedure: Pelvic lymph node dissection — Bilateral extended pelvic lymph node dissection
  Arms: Radical prostatectomy with an extended pelvic lymph node dissection

SUMMARY:
An extended pelvic lymph node dissection (ePLND) is the most accurate staging method to assess the presence of lymph node metastases in prostate cancer (PCa) patients. The therapeutic value, however remains unclear. Prospective randomized trials to address this void are lacking. Since in intermediate and a proportion of high risk PCa the risk of nodal metastases is generally below 25%, the vast majority of men undergo a procedure that has no oncological benefit, but is not without toxicity.

Therefore, the investigators aim to compare the oncologic outcomes of intermediate- and high-risk PCa patients with an estimated risk of lymph node invasion of 5-20% undergoing a radical prostatectomy (RP) with or without an ePLND.

DETAILED DESCRIPTION:
The role of an extended pelvic lymph node dissection (ePLND) in patients undergoing radical prostatectomy (RP) remains controversial. An ePLND is the most accurate staging method to assess the presence of lymph node metastases. Lymph node involvement is associated with a significantly worse prognosis and may require immediate or delayed adjuvant therapy. However, an ePLND is associated with an increased risk of complications such as lymphoceles, thromboses and lymphedema, and prolongs surgery and patient recovery. Thus, the diagnostic advantage of PLND should be weighed against the potential morbidity.

The therapeutic value of an ePLND remains especially unclear in PCa patients with an estimated risk of lymph node invasion (LNI) ≤ 20%, where only a minority of patients will have nodes harbouring metastases. Prospective trials to address this issue are still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥ 18 years
* Prostate cancer patients with a Briganti calculated risk of LN metastases of 5-20% without evidence of metastases on Prostate-Specific Membrane Antigen (PSMA) PET/CT requiring an ePLND in the standard treatment
* Scheduled for a (robot-assisted) laparoscopic radical prostatectomy
* Written informed consent

Exclusion Criteria:

* American Society of Anaesthesiology (ASA) classification > 3
* Patients with a contradiction for a lymphadenectomy
* Neoadjuvant hormone deprivation therapy
* Absence or withdrawal of an informed consent
* Evidence of metastases on pre-operative PSMA PET/CT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Presence of prostate cancer
Enrollment: 284 (Estimated)
Dates: Start 2021-11-17 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Persistent PSA rate | 6 months after surgery
  Persistent PSA is defined as a PSA value ≥ 0.1 ng/ml after radical prostatectomy

SECONDARY OUTCOMES:
Biochemical recurrence (BCR) rate | 3 years after surgery
  BCR is defined as a PSA value ≥ 0.2 ng/ml after radical prostatectomy
Metastasis-free survival | 3 years after surgery
  This is defined as the time between radical prostatectomy to development of metastasis
Incidence of complications after surgery | 3 and 6 months after surgery
  According to Clavien-Dindo classification
Incidence of salvage therapy after primary surgery | 3 years after surgery
  I.e., androgen deprivation therapy, radiation therapy or salvage lymph node dissection
Global Quality of life after surgery | 6, 12, 24 and 36 months after surgery
  Quality of life (QoL) will be assessed with the EORTC Core Quality of Life questionnaire's (QLQ-C30) global QoL scale ranging from 0 to 100, higher scores indicate better QoL
Health-related quality of life of patients with prostate cancer | 6, 12, 24 and 36 months after surgery
  Health-related quality of life in prostate cancer patients will be assessed with the EORTC Quality of Life Questionnaire - Prostate Cancer Module (QLQ-PR25) with a scale ranging from 0 to 100, higher scores indicate either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of (sexual) activity or functioning
Urinary continence after surgery | 6, 12, 24 and 36 months after surgery
  Urinary continence will be assessed with the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) questionnaire, ranging from 0 (best) to 21 (worst)
Urinary voiding symptoms | 6, 12, 24 and 36 months after surgery
  Urinary voiding symptoms will be assessed with the International Prostatic Symptoms Score (IPSS), ranging from 0 (best) to 35 (worst)
Potency after surgery | 6, 12, 24 and 36 months after surgery
  Potency will be assessed with the International Index of Erectile Function (IIEF) questionnaire. The IIEF classifies the severity of erectile dysfunction into five categories stratified by score:
  No erectile dysfunction. Score: 26-30 Mild erectile dysfunction. Score: 22-25 Mild to moderate erectile dysfunction. Score: 17-21 Moderate erectile dysfunction. Score: 11-16 Severe erectile dysfunction. Score: 6-10.

CONTACTS AND LOCATIONS:
Overall Officials: Henk G van der Poel, Prof, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No